CLINICAL TRIAL: NCT04810286
Title: Comparison of Prefabricated Myofunctional Appliances and 3D-Printing Myofunctional Appliances in Children With Class II Division 1 Malocclusion
Brief Title: Prefabricated Versus 3D-Printing Myofunctional Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Suleyman Kutalmış Buyuk, Associate Professor Dr., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-47
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Myofunctional treatment; 3D-Print; Prefabricated myofunctional appliance; Class II division 1 malocclusion; Orthodontics
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 3D-print myofunctional appliance
  Interventions: Procedure: 3d-Printing Myofunctional Appliance
- Control Group (Active Comparator): Prefabricated myfunctional appliance
  Interventions: Procedure: 3d-Printing Myofunctional Appliance

INTERVENTIONS:
Procedure: 3d-Printing Myofunctional Appliance — To evaluate soft- and hard-tissue changes Class II division 1 tchildren with a prefabricated myofunctional appliance versus a 3D-printed myofunctional appliance.

SUMMARY:
The aim of this clinical study is to evaluate the dentoskeletal effects of Class II division 1 treatment in growing patients with a prefabricated myofunctional appliance versus a 3D-printing myofunctional appliance.

DETAILED DESCRIPTION:
This study aims to investigate the dentoskeletal effects of Class II division 1 treatment in growing patients with a prefabricated myofunctional appliance versus a 3D-printing myofunctional appliance.

ELIGIBILITY:
Inclusion Criteria:

* Increased overjet >4 mm
* Skeletal Class II relationship (ANB > 4 degree)
* No previous orthodontic treatment

Exclusion Criteria:

-Craniofacial syndrome

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of dentoskeletal changes | 1 year
  Dentoskeletal effects of appliances

CONTACTS AND LOCATIONS:
Overall Officials: Suleyman Kutalmış Buyuk, PhD, Study Chair — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No